CLINICAL TRIAL: NCT00174993
Title: PROspective PioglitAzone Clinical Trial In MacroVascular Events: A Macrovascular Outcome Study in Type 2 Diabetic Patients Comparing Pioglitazone With Placebo in Addition to Existing Therapy
Brief Title: Efficacy of Pioglitazone on Macrovascular Outcome in Patients With Type 2 Diabetes
Acronym: PROactive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD4833/EC444; U1111-1114-2854 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone QD (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15 mg to 45 mg, tablets, orally, once daily for up to 48 months.
  Other Names: Actos; AD4833
  Arms: Pioglitazone QD
Drug: Placebo — Pioglitazone placebo-matching tablets, orally, once daily for up to 48 months
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine whether pioglitazone, once daily (QD), can delay the time to death, heart attack, acute coronary syndrome, heart bypass surgery, stroke, leg bypass surgery or amputation in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Diabetes mellitus is one of the most common non-communicable diseases worldwide. More than 22 million persons have been diagnosed with diabetes in the European region of the International Diabetes Federation. Complications of diabetes involving both microvascular and macrovascular systems contribute to increased disability and reduced life expectancy. Damage to the coronary, cerebral (brain), and peripheral vascular beds as a consequence of diabetes is responsible for the increased macrovascular illness and death associated with the disease.

Insulin resistance is common to the genesis of both atherosclerosis and type 2 diabetes mellitus. In diabetes, insulin resistance is coupled to receptor dysfunction. In atherosclerosis, insulin resistance may have both direct effects on the cardiovascular system as well as indirect effects provoked by imbalances in blood glucose, lipids, clotting factors, endothelial function, and other factors. Considerable indirect evidence suggests that peroxisome proliferator-activated receptor agonists may favorably influence macrovascular outcome, either through modification of risk factors (such as blood lipids) or through effects on the vessel wall.

Pioglitazone, a thiazolidinedione compound discovered by Takeda Pharmaceutical Company, Ltd, functions as a peroxisome proliferator-activated receptor agonist as its mode of action.

This study is designed to assess whether pioglitazone in combination with other medications administered for glycemic management of type 2 diabetes might reduce the incidence of macrovascular events associated with this disease compared with placebo. Individuals who participate in this study will provide written informed consent and will be required to commit to screening and randomization visits and approximately 17 additional visits (1 every 2 months for the first year and every 3 months thereafter) at the study center. Study participation is anticipated to be about 40 months (or approximately 3 years and 4 months). Multiple procedures will occur at each visit which may include fasting, blood collection, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria

* Type 2 diabetes mellitus
* Glycosylated hemoglobin above the upper limit of normal (ie, the local equivalent of 6.5% for)
* Established history of macrovascular disease, defined as 1 or more of:

  * Myocardial infarction at least 6 months before entry into the study.
  * Stroke at least 6 months before entry into the study
  * Percutaneous coronary intervention or coronary artery bypass graft at least 6 months before entry into the study.
  * Acute coronary syndrome at least 3 months before entry into the study.
  * Objective evidence of coronary artery disease.
  * Peripheral arterial obstructive disease

Exclusion Criteria

* Signs of type 1 diabetes.
* Patients prescribed insulin as sole therapy for glycemic control of diabetes for 2 weeks or more at any time in the previous 3 months.
* Myocardial infarction, stroke, coronary artery bypass graft, or percutaneous cardiac intervention in the 6 months prior to enrolment.
* Acute coronary syndrome in the 3 months prior to enrolment.
* Heart failure at entry defined as patient having a New York Heart Association functional score of II or above.
* Had an appointment for a coronary angiogram or endovascular or surgical intervention.
* Leg ulcers, gangrene, or ischemic rest pain.
* Had an appointment for an angiogram or endovascular or surgical intervention for leg ischemia.
* Had undergone a major operation (defined as a surgical procedure lasting for more than 30 minutes) at any time in the previous 4 weeks.
* Significantly impaired hepatic function, defined as alanine aminotransferase greater than 2.5 times the upper limit of normal.
* Familial polyposis coli.
* Required dialysis.
* History of alcohol or drug abuse.
* Any other intercurrent disease believed to be likely to have a significant impact on the patient's life expectancy during the course of the study (eg, cancer).
* Patient was undergoing follow-up as part of another clinical trial or less than 3 months had elapsed since the last dose of an investigational drug or procedure.
* Hypersensitivity to pioglitazone or other TZD.
* Current use of pioglitazone or other TZD.
* Patient was known to be infected with human immunodeficiency virus or was known to have viral hepatitis.
* Women who were any of the following: pregnant, breast feeding, wished to become pregnant during the course of the study or of childbearing potential and not planning to use a reliable method of contraception throughout the study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4373 (Actual)
Dates: Start 2001-05; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Time to the Composite of All Cause Mortality, Non-Fatal Myocardial Infarction, Stroke, Acute Coronary Syndrome, Major Leg Amputation, Cardiac Intervention, Bypass Surgery or Leg Revascularization. | At First Occurrence

SECONDARY OUTCOMES:
Time to All Cause Mortality. | At occurrence
Time to Non-Fatal Myocardial Infarction. | At occurrence
Time to Acute Coronary Syndrome. | At occurrence
Time to Cardiac Intervention (including coronary artery bypass graft or percutaneous coronary intervention). | At occurrence
Time to Stroke. | At occurrence
Time to Major Leg Amputation (above the ankle). | At occurrence
Time to Bypass Surgery | At occurrence
Time to Revascularization of the Leg. | At occurrence
Time to Cardiovascular Mortality. | At occurrence

CONTACTS AND LOCATIONS:
Overall Officials: European Development Director, Study Director — Takeda
Locations (19):
- Multiple Cities, Austria
- Multiple Cities, Belgium
- Multiple Cities, Czechia
- Multiple Cities, Denmark
- Multiple Cities, Estonia
- Multiple Cities, Finland
- Multiple Cities, France
- Multiple Cities, Germany
- Multiple Cities, Hungary
- Multiple Cities, Italy
- Multiple Cities, Latvia
- Multiple Cities, Lithuania
- Multiple Cities, Netherlands
- Multiple Cities, Norway
- Multiple Cities, Poland
- Multiple Cities, Slovakia
- Multiple Cities, Sweden
- Multiple Cities, Switzerland
- Multiple Cities, United Kingdom

REFERENCES:
- [Background] Bottomley JM, Palmer AJ, Williams R, Dormandy JA, Massi-Benedetti M. PROactive 03: Pioglitazone, type 2 diabetes and reducing macrovascular events - economic implications?. Br J Diabetes Vasc Dis 2006;6(Pt 2):64-69
- [Background] Kirby,M, Heart Disease Prevention - What Place for the Glitazones. Br J Cardiol 2006;13:(1):66-70.
- [Background] Brandle M, Goodall G, Erny-Albrecht KM, Erdmann E, Valentine WJ. Cost-effectiveness of pioglitazone in patients with type 2 diabetes and a history of macrovascular disease in a Swiss setting. Swiss Med Wkly. 2009 Mar 21;139(11-12):173-84. doi: 10.4414/smw.2009.12381. PMID 19330561
- [Background] Betteridge DJ, DeFronzo RA, Chilton RJ. PROactive: time for a critical appraisal. Eur Heart J. 2008 Apr;29(8):969-83. doi: 10.1093/eurheartj/ehn114. Epub 2008 Mar 28. PMID 18375395
- [Background] Scherbaum WA, Goodall G, Erny-Albrecht KM, Massi-Benedetti M, Erdmann E, Valentine WJ. Cost-effectiveness of pioglitazone in type 2 diabetes patients with a history of macrovascular disease: a German perspective. Cost Eff Resour Alloc. 2009 May 5;7:9. doi: 10.1186/1478-7547-7-9. PMID 19416529
- [Background] van Troostenburg de Bruyn AR, Dormandy J. Risk of thiazolidinedione-associated fracture should be appropriately assessed. Arch Intern Med. 2010 Jan 25;170(2):209-10. doi: 10.1001/archinternmed.2009.487. No abstract available. PMID 20101019
- [Result] Dormandy JA, Charbonnel B, Eckland DJ, Erdmann E, Massi-Benedetti M, Moules IK, Skene AM, Tan MH, Lefebvre PJ, Murray GD, Standl E, Wilcox RG, Wilhelmsen L, Betteridge J, Birkeland K, Golay A, Heine RJ, Koranyi L, Laakso M, Mokan M, Norkus A, Pirags V, Podar T, Scheen A, Scherbaum W, Schernthaner G, Schmitz O, Skrha J, Smith U, Taton J; PROactive Investigators. Secondary prevention of macrovascular events in patients with type 2 diabetes in the PROactive Study (PROspective pioglitAzone Clinical Trial In macroVascular Events): a randomised controlled trial. Lancet. 2005 Oct 8;366(9493):1279-89. doi: 10.1016/S0140-6736(05)67528-9. PMID 16214598
- [Result] Schneider CA, Ferrannini E, Defronzo R, Schernthaner G, Yates J, Erdmann E. Effect of pioglitazone on cardiovascular outcome in diabetes and chronic kidney disease. J Am Soc Nephrol. 2008 Jan;19(1):182-7. doi: 10.1681/ASN.2007060678. Epub 2007 Dec 5. PMID 18057215
- [Result] Ryden L, Thrainsdottir I, Swedberg K. Adjudication of serious heart failure in patients from PROactive. Lancet. 2007 Jan 20;369(9557):189-90. doi: 10.1016/S0140-6736(07)60106-8. No abstract available. PMID 17240282
- [Result] Erdmann E, Dormandy J, Wilcox R, Massi-Benedetti M, Charbonnel B. PROactive 07: pioglitazone in the treatment of type 2 diabetes: results of the PROactive study. Vasc Health Risk Manag. 2007;3(4):355-70. PMID 17969365
- [Result] Erdmann E, Dormandy JA. The Effect of Pioglitazone on Recurrent Myocardial Infarction in 2445 Patients with Type 2 Diabetes and Preexisting Myocardial Infarction - Data from the PROactive Study. Circulation 2005;112:(21):3364-3364
- [Result] Erdmann E, Dormandy JA, Charbonnel B, Massi-Benedetti M, Moules IK, Skene AM; PROactive Investigators. The effect of pioglitazone on recurrent myocardial infarction in 2,445 patients with type 2 diabetes and previous myocardial infarction: results from the PROactive (PROactive 05) Study. J Am Coll Cardiol. 2007 May 1;49(17):1772-80. doi: 10.1016/j.jacc.2006.12.048. Epub 2007 Apr 16. PMID 17466227
- [Result] Valentine WJ, Bottomley JM, Palmer AJ, Brandle M, Foos V, Williams R, Dormandy JA, Yates J, Tan MH, Massi-Benedetti M; PROactive Study Group. PROactive 06: cost-effectiveness of pioglitazone in Type 2 diabetes in the UK. Diabet Med. 2007 Sep;24(9):982-1002. doi: 10.1111/j.1464-5491.2007.02188.x. Epub 2007 Jun 25. PMID 17593245
- [Result] Wilcox R, Bousser MG, Betteridge DJ, Schernthaner G, Pirags V, Kupfer S, Dormandy J; PROactive Investigators. Effects of pioglitazone in patients with type 2 diabetes with or without previous stroke: results from PROactive (PROspective pioglitAzone Clinical Trial In macroVascular Events 04). Stroke. 2007 Mar;38(3):865-73. doi: 10.1161/01.STR.0000257974.06317.49. Epub 2007 Feb 8. PMID 17290029
- [Result] Erdmann E, Charbonnel B, Wilcox RG, Skene AM, Massi-Benedetti M, Yates J, Tan M, Spanheimer R, Standl E, Dormandy JA; PROactive Investigators. Pioglitazone use and heart failure in patients with type 2 diabetes and preexisting cardiovascular disease: data from the PROactive study (PROactive 08). Diabetes Care. 2007 Nov;30(11):2773-8. doi: 10.2337/dc07-0717. Epub 2007 Jul 31. PMID 17666462
- [Result] Valentine WJ, Tucker D, Palmer AJ, Minshall ME, Foos V, Silberman C; PROactive Study Group. Long-term cost-effectiveness of pioglitazone versus placebo in addition to existing diabetes treatment: a US analysis based on PROactive. Value Health. 2009 Jan-Feb;12(1):1-9. doi: 10.1111/j.1524-4733.2008.00403.x. Epub 2008 Jul 24. PMID 18657104
- [Result] Wilcox R, Kupfer S, Erdmann E; PROactive Study investigators. Effects of pioglitazone on major adverse cardiovascular events in high-risk patients with type 2 diabetes: results from PROspective pioglitAzone Clinical Trial In macro Vascular Events (PROactive 10). Am Heart J. 2008 Apr;155(4):712-7. doi: 10.1016/j.ahj.2007.11.029. Epub 2008 Feb 21. PMID 18371481
- [Result] Charbonnel B, Dormandy J, Erdmann E, Massi-Benedetti M, Skene A; PROactive Study Group. The prospective pioglitazone clinical trial in macrovascular events (PROactive): can pioglitazone reduce cardiovascular events in diabetes? Study design and baseline characteristics of 5238 patients. Diabetes Care. 2004 Jul;27(7):1647-53. doi: 10.2337/diacare.27.7.1647. PMID 15220241
- [Result] Spanheimer R, Betteridge DJ, Tan MH, Ferrannini E, Charbonnel B; PROactive Investigators. Long-term lipid effects of pioglitazone by baseline anti-hyperglycemia medication therapy and statin use from the PROactive experience (PROactive 14). Am J Cardiol. 2009 Jul 15;104(2):234-9. doi: 10.1016/j.amjcard.2009.03.023. Epub 2009 Jun 3. PMID 19576353
- [Result] Scheen AJ, Tan MH, Betteridge DJ, Birkeland K, Schmitz O, Charbonnel B; PROactive investigators. Long-term glycaemic control with metformin-sulphonylurea-pioglitazone triple therapy in PROactive (PROactive 17). Diabet Med. 2009 Oct;26(10):1033-9. doi: 10.1111/j.1464-5491.2009.02816.x. PMID 19900236
- [Result] Scheen AJ, Tan MH, Betteridge DJ, Birkeland K, Schmitz O, Charbonnel B; PROactive investigators. Long-term glycaemic effects of pioglitazone compared with placebo as add-on treatment to metformin or sulphonylurea monotherapy in PROactive (PROactive 18). Diabet Med. 2009 Dec;26(12):1242-9. doi: 10.1111/j.1464-5491.2009.02857.x. PMID 20002476
- [Result] Dormandy JA, Betteridge DJ, Schernthaner G, Pirags V, Norgren L; PROactive investigators. Impact of peripheral arterial disease in patients with diabetes--results from PROactive (PROactive 11). Atherosclerosis. 2009 Jan;202(1):272-81. doi: 10.1016/j.atherosclerosis.2008.03.002. Epub 2008 Mar 18. PMID 18538774
- [Result] Spanheimer,RG, Ferrannini,E, Long term effects of pioglitazone on diabetic dyslipidemia independent of baseline statin use and antihyperglycemic medication: a review from PROactive. Asia Pac J Cardiol 2009;1:(1):75-81.
- [Result] Dormandy J, Bhattacharya M, van Troostenburg de Bruyn AR; PROactive investigators. Safety and tolerability of pioglitazone in high-risk patients with type 2 diabetes: an overview of data from PROactive. Drug Saf. 2009;32(3):187-202. doi: 10.2165/00002018-200932030-00002. PMID 19338377
- [Result] Betteridge DJ. CHICAGO, PERISCOPE and PROactive: CV risk modification in diabetes with pioglitazone. Fundam Clin Pharmacol. 2009 Dec;23(6):675-9. doi: 10.1111/j.1472-8206.2009.00741.x. Epub 2009 Sep 10. PMID 19744248
- [Result] Erdmann E, Spanheimer R, Charbonnel B; PROactive Study Investigators. Pioglitazone and the risk of cardiovascular events in patients with Type 2 diabetes receiving concomitant treatment with nitrates, renin-angiotensin system blockers, or insulin: results from the PROactive study (PROactive 20). J Diabetes. 2010 Sep;2(3):212-20. doi: 10.1111/j.1753-0407.2010.00082.x. PMID 20923486
- [Result] Ferrannini E, Betteridge DJ, Dormandy JA, Charbonnel B, Wilcox RG, Spanheimer R, Erdmann E, Defronzo RA, Laakso M. High-density lipoprotein-cholesterol and not HbA1c was directly related to cardiovascular outcome in PROactive. Diabetes Obes Metab. 2011 Aug;13(8):759-64. doi: 10.1111/j.1463-1326.2011.01404.x. PMID 21457426
- [Derived] Doehner W, Erdmann E, Cairns R, Clark AL, Dormandy JA, Ferrannini E, Anker SD. Inverse relation of body weight and weight change with mortality and morbidity in patients with type 2 diabetes and cardiovascular co-morbidity: an analysis of the PROactive study population. Int J Cardiol. 2012 Dec 15;162(1):20-6. doi: 10.1016/j.ijcard.2011.09.039. Epub 2011 Oct 29. PMID 22037349
- [Derived] Pfister R, Cairns R, Erdmann E, Schneider CA; PROactive investigators. Prognostic impact of electrocardiographic signs in patients with Type 2 diabetes and cardiovascular disease: results from the PROactive study. Diabet Med. 2011 Oct;28(10):1206-12. doi: 10.1111/j.1464-5491.2011.03281.x. PMID 21388447
- [Derived] Charbonnel B, DeFronzo R, Davidson J, Schmitz O, Birkeland K, Pirags V, Scheen A; PROactive investigators. Pioglitazone use in combination with insulin in the prospective pioglitazone clinical trial in macrovascular events study (PROactive19). J Clin Endocrinol Metab. 2010 May;95(5):2163-71. doi: 10.1210/jc.2009-1974. Epub 2010 Mar 17. PMID 20237169
- See also: ACTOS Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI